CLINICAL TRIAL: NCT00668317
Title: An 8 Week Non-selected Cohort Study to Investigate Whether the Treatment of Reflux Induced Cough Alters Associated Bronchial Hyper-responsiveness
Brief Title: Bronchial Hyper-responsiveness in Reflux Cough
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Primary care physicians began prescribing antacid therapy for chronic cough
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2006-004102-13
Record Dates: First submitted 2008-04-24; First posted 2008-04-29 (Estimated); Results first posted 2012-11-16 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Cough
Keywords: Hyper-responsiveness, reflux cough
MeSH Terms: conditions — Cough | interventions — Omeprazole; Ranitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- omeprazole and ranitidine (Other): 20 mg oralomeprazole oral tablet twice daily and ranitidine 300 mg oral tablet once daily nocte
  Interventions: Drug: Omeprazole; Drug: Ranitidine

INTERVENTIONS:
Drug: Omeprazole — 20 mg BD tablet 8 weeks duration
  Other Names: Losec
Drug: Ranitidine — 300 mg od nocte tablet 8weeks duration
  Other Names: Zantac

SUMMARY:
The study aim is to determine the effect of 8 weeks of anti-reflux treatment (full acid suppression) on bronchial hyper-responsiveness and whether there is a symptomatic improvement.

ELIGIBILITY:
Inclusion Criteria:

* Positive methacholine challenge test PC20 less than 4mg/ml (Can be previously documented in patients notes within last 4weeks)
* Written informed consent
* Patients with a history of chronic cough (at least 3 months duration), and associated symptoms of gastro-oesophageal reflux
* Male and female subjects of at least 18 yrs of age
* Subjects able to perform satisfactory FEV1 manoeuvres
* Subjects able to understand the study and co-operate with the study procedures
* Subjects who consent to their general practitioner (GP) being informed of their study participation

Exclusion Criteria:

* has had a heart attack in the last three months
* suffers from angina, hypertension or ischaemic heart disease
* has epilepsy for which he/she is taking medication
* FEV1< 60% predicted
* FEV1<1.6L
* Female subjects who are pregnant, or lactating, or who are of child bearing potential but are not using contraceptive measures
* Suffering from any concomitant disease which may interfere with study procedures or evaluation.
* A lower respiratory tract infection 4 weeks prior to entry on to study
* Participation in another study (use of investigational product) within 30 days preceding entry on to study.
* Alcohol or drug abuse
* Use of opiates to treat cough 1 week prior to enrollment
* Subjects who are taking Angiotensin Converting Enzymes (ACE) inhibitors.
* Subjects who have significant pathology on most recent chest X-Ray.
* Inability to understand the procedures and the implications of a challenge test
* Patients already taking or have taken in last 4 weeks PPI and H2 receptor antagonist (full acid suppression treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2006-09; Primary Completion 2009-09 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alyn H Morice, Professor, Principal Investigator — Hull University Teaching Hospitals NHS Trust
Locations (1):
- Clinical Trials Unit , Cardiovascular and respiratory studies, Castle Hill Hospital, Cottingham, East Yorkshire, United Kingdom

REFERENCES:
- [Background] Morice AH, Kastelik JA, Thompson R. Cough challenge in the assessment of cough reflex. Br J Clin Pharmacol. 2001 Oct;52(4):365-75. doi: 10.1046/j.0306-5251.2001.01475.x. No abstract available. PMID 11678780
- See also: Publication Link — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC2014577/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited at the cough clinic at castleHill Hospital
Pre-assignment Details: Patients had to have a positive methacholine challenge, and reflux associated chronic cough
Groups:
- Antacid Therapy: Therapy with omeprazole 20 mg BD and Ranitidine 300mg od nocte
Period: Overall Study
Arm/Group | Antacid Therapy
Started | 5
Completed | 3
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Arm/Group | Antacid Therapy
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.8 (8.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 1
Region of Enrollment [Number; unit: participants]
  United Kingdom | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Methacholine Sensitivity
Description: Concentration of methacholine (mg/ml) at which participants forced expired volume in 1 sec (FEV1) is reduced by 20% (the provocation concentration of methacholine causing a 20% fall in FEV1-PC20).
  To measure if there is a significant difference in PC20 recorded at baseline to that recorded following 8 weeks treatment with omeprazole and ranitidine
Time Frame: baseline and 8 weeks
Population: All subjects recruited with efficacy data recorded after week T0 will be included in the ITT population for analysis. Assuming a within subject standard deviation(for change in PC20) of no more than 2.71 units, 30 subjects are sufficient to provide 80% power to detect a treatment difference of 1.8 units using a 5% two sided significance test
Measure: Mean (Standard Deviation); unit: mg/ml
Groups:
- Omeprazole and Ranitidine: Therapy with omeprazole 20 mg twice a day (BD) and Ranitidine 300mg once a day (od) at night (nocte)
Arm/Group | Omeprazole and Ranitidine
Number analyzed (Participants) | 3
mg/ml | 0.598 (0.479)

2. Secondary Outcome: Improvement in Cough Symptoms Measured Using Leicester Cough Questionnaire
Time Frame: 8 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 8 week
Description: data collected at each visit of the study
Arm/Group | Antacid Therapy
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes